CLINICAL TRIAL: NCT05697120
Title: Effect of Using a Smartphone Application to Promote Adherence to Healthy Behaviour Post-cardiac Rehabilitation: Five Year Follow-up of a Randomized Controlled Trial
Brief Title: Long-term Effects of Individualized Follow-up With an App for One Year
Status: Completed | Type: Observational
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Sponsor
Other Study IDs: OsloMetU
Record Dates: First submitted 2022-11-03; First posted 2023-01-25 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease
Keywords: Cardiac rehabilitation; mHealth; mobile phone app; Lifestyle; Smartphone
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to examine the long-term (3-5 year post intervention) effects post individualized follow-up with an app for one year, compared to a control group that received usual care on factors related to healthy behaviour in patients post-CR.

DETAILED DESCRIPTION:
Recently, our research group demonstrated that individualized follow-up with an app for one year post-Cardiac Rehabilitation (post-CR) significantly improved exercise capacity, exercise habits and self-perceived goal achievement compared to a control group receiving usual care. To prepare for real-world implementation of an app to promote healthy behaviour post-CR, we will investigate the long-term effects (3-5 year post intervention). The aim of this study is to examine the long-term (3-5 year post intervention) effects post individualized follow-up with an app for one year, compared to a control group that received usual care on factors related to healthy behaviour in patients post-CR. We hypothesize that patients allocated to the intervention group post-CR have internalized healthy behaviour and therefore have significantly higher exercise capacity and lower bodyweight compared to the control group, 3-5year post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Included in the RCT of which this study is built on

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients participating in cardiac rehabilitation. The sample in this study will be the same as in the RCT of which this study is built on (ClinicalTrials.gov NCT03174106)
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake | 5 year post rehab
  Relative VO2peak (ml/kg/min)

SECONDARY OUTCOMES:
Time to exhaustion | 5 year post rehab
  Time on treadmill measured in seconds
Peak incline | 5 year post rehab
  Incline (%) at treadmill in the end of the test
Peak velocity | 5 year post rehab
  Kilometer per hour in the end of the test
Bodyweight | 5 year post rehab
  Kilograms
LDL cholesterol | 5 year post rehab
  Blood sample
HDL cholesterol | 5 year post rehab
  Blood sample
Total cholesterol | 5 year post rehab
  Blood sample
Exercise habits | 5 year post rehab
  Mean number of exercise sessions each week for the last year
Health related quality of life | 5 year post rehab
  HeartQoL
Health status | 5 year post rehab
  EQ5D
Cardiovascular events | 5 year post rehab
  Number of new cardiovascular events in the last five years
Dietary habits | 5 year post rehab
  "Hva spiser du" - a norwegian questionnaire developed to assess nutrional habits
Triglycerides | 5 year post rehab
  Bloodsample
Physical activity | 5 year post rehab
  IPAQ

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo Metropolitan University, Oslo, Norway

REFERENCES:
- [Derived] Lunde P, Bye A, Grimsmo J, Pripp AH, Ritschel V, Jarstad E, Nilsson BB. Effects of Individualized Follow-Up With an App Postcardiac Rehabilitation: Five-Year Follow-Up of a Randomized Controlled Trial. J Med Internet Res. 2025 Feb 13;27:e60256. doi: 10.2196/60256. PMID 39946716

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT05697120/SAP_000.pdf